CLINICAL TRIAL: NCT02597478
Title: A Preliminary Study of Prophylactic Fentanyl Sublingual Spray for Exercise-Induced Breakthrough Dyspnea
Brief Title: Fentanyl Sublingual Spray for Exercise-Induced Breakthrough Dyspnea
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-0137; NCI-2015-02132 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Results first posted 2020-12-08 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Fentanyl Sublingual Spray; Fentanyl SL Spray; FSS; Questionnaires; Surveys; Mental Abilities Test; Phone Call; Shuttle Walk Test
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low-Dose Fentanyl Spray Group (Experimental): Questionnaires completed at baseline and at end of study visit. Participant performs Shuttle Walk Test before and after receiving low-dose Fentanyl sublingual spray. Four mental ability tests completed after each walk test. Low-dose Fentanyl sprayed into mouth and under tongue one hour after first Shuttle Walk Test.
  Interventions: Drug: Fentanyl Sublingual Spray; Procedure: Shuttle Walk Test; Behavioral: Questionnaires; Behavioral: Mental Ability Tests; Behavioral: Phone Call
- High-Dose Fentanyl Spray Group (Experimental): Questionnaires completed at baseline and at end of study visit. Participant performs Shuttle Walk Test before and after receiving high-dose Fentanyl sublingual spray. Four mental ability tests completed after each walk test. High-dose Fentanyl sprayed into mouth and under tongue one hour after first Shuttle Walk Test.
  Interventions: Drug: Fentanyl Sublingual Spray; Procedure: Shuttle Walk Test; Behavioral: Questionnaires; Behavioral: Mental Ability Tests; Behavioral: Phone Call

INTERVENTIONS:
Drug: Fentanyl Sublingual Spray — Low-dose Fentanyl Goup: 15-25% of the morphine equivalent daily dose (MEDD) sprayed into mouth and under tongue one hour after first Shuttle Walk Test.
  High-Dose Fentanyl Group: 35-45% of the morphine equivalent daily dose (MEDD) sprayed into mouth and under tongue one hour after first Shuttle Walk Test.
  Other Names: Fentanyl SL Spray; FSS
Procedure: Shuttle Walk Test — Participants walk back and forth between 2 cones in an indoor hallway for up to 12 minutes. After one hour Fentanyl Spray delivered, then second walk test performed.
Behavioral: Questionnaires — Questionnaire completed about any breathing problems or other symptoms participant may be having at baseline. End of study questionnaire asks which dose level of study drug participant thinks they received. Participant also completes a questionnaire about how study drug may have helped them and how satisfied they are with the study. It should take about 5 minutes to complete the questionnaire.
  Other Names: Surveys
Behavioral: Mental Ability Tests — After each walk test, participant completes 4 tests of their mental abilities. It should take 15 minutes total to complete these tests.
Behavioral: Phone Call — Thirty days study visit participant called by study staff. This call should last about 10 minutes.

SUMMARY:
The goal of this clinical research study is to learn if fentanyl can help shortness of breath in cancer patients. Researchers also want to learn if the study drug can help to improve your physical function.

DETAILED DESCRIPTION:
If you agree to take part in this study, the study staff will collect information from your medical record about your age, sex, race, and disease type, as well as how well you are able to perform the normal activities of daily living, any drugs you are taking, and any possible causes of shortness of breath.

Study Groups:

You will be randomly assigned (as in the flip of a coin) to receive either low-dose or high-dose fentanyl spray. This is done because no one knows if one study group is better, the same, or worse than the other group.

Study Visit:

During your study visit, you will complete 2 questionnaires about any breathing problems or other symptoms you may be having. It should take about 10 minutes total to complete these questionnaires.

You will blow into a device called a spirometer a few times to measure your lung function. You will also be asked to inhale into another device called a negative inspiratory force meter (NIF). This device measures the volume of air that can be inhaled after normal breathing.

The study staff will then record your vital signs (heart rate, breathing rate, blood pressure, and your blood-oxygen level). Your blood-oxygen level will be measured with a device that will be clipped gently onto your fingertip). You will then be asked how hard it is to catch your breath and to rate your level of tiredness.

When instructed, you will walk back and forth between 2 cones in an indoor hallway for up to 12 minutes. This is called the Shuttle Walk Test. The purpose of this timed test is to see how far and fast you can walk without stopping for a rest. You will be asked to pivot briskly around the cones and continue back the other way. You may stop this test at any time if you feel you cannot continue.

After that, you will sit down and rest for up to 1 hour. During this time, the study drug will be prepared, and you may be asked at different times how hard it is to catch your breath.

After the rest period, you will be given the fentanyl to spray into your mouth and under your tongue. About 10 minutes later, you will be asked about any side effects you may be having.

At that point, you will perform a second Shuttle Walk Test. Then the study staff will ask you again about any side effects you may be having, your level of tiredness, and how hard it is to catch your breath. Your vital signs will also be measured. The total distance you walked will also be recorded.

After each walk test, you will also be asked to complete 4 tests of your mental abilities, including finger tapping, simple math questions (addition, subtraction, multiplication, division), recall of numbers, and recall of objects. It should take 15 minutes total to complete these tests.

At the end of the study visit, you will be asked which dose level of the study drug you think you received (high-dose or low-dose). You will also complete a questionnaire about how the study drug may have helped you and how satisfied you are with the study. It should take about 5 minutes to complete the questionnaire.

At the end of the study, if you think that taking fentanyl helped to improve your breathing, your doctor will be told, so that you and your doctor may discuss if fentanyl would be helpful to you in the future.

Length of Study:

Your active participation in this study is over after you complete the last questionnaire. You will be taken off study if intolerable side effects occur or if you are unable to follow study directions.

Follow-Up:

Fourteen (14) days after your study visit you will be called by the study staff and asked how you are feeling and about any side effects you may be having. This call should last about 10 minutes.

This is an investigational study. Fentanyl is FDA approved and commercially available for the treatment of pain. Its use to control shortness of breath is investigational.

Up to 30 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cancer with evidence of active disease
2. Breakthrough dyspnea, defined as dyspnea with an average intensity level over the past 7 days of at least 3/10 on a numeric rating scale upon significant exertion or continuous dyspnea </=7/10 with worsening upon significant exertion
3. Outpatient at MD Anderson Cancer Center seen by the Supportive Care Service, Thoracic Medical Oncology, Cancer Pain Clinic, or Cardiopulmonary clinic
4. Ambulatory and able to walk with or without walking aid
5. On strong opioids with morphine equivalent daily dose of 80-500 mg for at least one week, with stable (i.e. +/- 30%) regular dose over the last 24 hours
6. Karnofsky performance status >/=50%
7. Age 18 or older
8. Able to complete study assessments

Exclusion Criteria:

1. Dyspnea at rest >/=7/10 at the time of enrollment
2. Supplemental oxygen requirement >6 L per minute
3. Delirium (i.e. Memorial delirium rating scale >13)
4. History of unstable angina or myocardial infarction 1 month prior to study enrollment
5. Resting heart rate >120 at the time of study enrollment
6. Systolic pressure >180 mmHg or diastolic pressure >100 mmHg at the time of study enrollment
7. History of active opioid abuse within the past 12 months
8. History of allergy to fentanyl
9. Severe anemia (Hb <7g/L) if documented in the last month and not corrected prior to study enrollment*
10. Diagnosis of acute pulmonary embolism within past 2 weeks
11. Diagnosis of pulmonary hypertension
12. Unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2021-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants (age>18) with an active diagnosis of cancer were recruited between 1/2016 and 10/2018 from the Supportive Care and Thoracic Medical Oncology outpatient clinics at MD Anderson Cancer Center who met the inclusion and exclusion criteria.
Pre-assignment Details: A total of 50 participants enrolled but 34 patients were randomized to start the study. 13 became symptomatic while on wait list and could not proceed, 2 participants died, and 1 had screen failure before participants were randomized.
Groups:
- Intervention Group (High Dose Fentanyl Sublingual Spray): Received Fentanyl sublingual spray 10 minutes before performing second shuttle walk test, dose was 35-45% of morphine equivalent daily dose.
- Controlled Group (Low Dose Fentanyl Sublingual Spray): Received Fentanyl sublingual spray 10 minutes before performing second shuttle walk test, dose was 15-20% of morphine equivalent daily dose.
Period: Overall Study
Arm/Group | Intervention Group (High Dose Fentanyl Sublingual Spray) | Controlled Group (Low Dose Fentanyl Sublingual Spray)
Started | 16 | 18
Completed | 13 | 17
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Change of opioid dose | 1 | 0
Not completed — Insufficient exertional dyspnea | 0 | 1

BASELINE CHARACTERISTICS:
Population: The data is provided for 30 participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group (High Dose Fentanyl Sublingual Spray) | Controlled Group (Low Dose Fentanyl Sublingual Spray) | Total
Number analyzed (Participants) | 13 | 17 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (16) | 51 (10) | 52 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 11 | 14 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 15 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 17 | 30
Education [Count of Participants; unit: Participants]
  High school or less | 7 | 2 | 9
  College | 6 | 12 | 18
  Advanced degree | 0 | 3 | 3
Cancer Type [Count of Participants; unit: Participants]
  Breast | 2 | 6 | 8
  Genitourinary | 2 | 2 | 4
  Gastrointestinal | 3 | 2 | 5
  Gynecological | 2 | 1 | 3
  Head and Neck | 0 | 2 | 2
  Respiratory | 4 | 3 | 7
  Others | 0 | 1 | 1
Cancer Stage [Count of Participants; unit: Participants]
  Metastatic or recurrent | 10 | 14 | 24
  Locally advanced | 3 | 2 | 5
  Localized | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Modified Dyspnea Borg Scale (Dyspnea Intensity)
Description: The primary outcome was dyspnea intensity "now" using the modified Borg scale, which ranges from 0 ("no shortness of breath") to 10 ("worst possible shortness of breath"). We measured the change in modified dyspnea Borg scale (0-10) between the first and second shuttle walk tests. This scale has been validated in multiple studies, with a minimal clinically significant difference of 1 point.
Time Frame: Before and after the first and second shuttle walk tests
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group (High Dose Fentanyl Sublingual Spray) | Controlled Group (Low Dose Fentanyl Sublingual Spray)
Number analyzed (Participants) | 13 | 17
score on a scale | -1.4 [-2.4 to -0.5] | -0.5 [-1.3 to 0.3]

2. Secondary Outcome: Modified Dyspnea Borg Scale (Dyspnea Unpleasantness)
Description: The modified Borg scale (dyspnea unpleasantness), which ranges from 0 ("no shortness of breath") to 10 ("worst possible shortness of breath"). We measured the change in modified dyspnea Borg scale (0-10) between the first and second shuttle walk tests.
Time Frame: Before and after the first and second shuttle walk tests
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group (High Dose Fentanyl Sublingual Spray) | Controlled Group (Low Dose Fentanyl Sublingual Spray)
Number analyzed (Participants) | 13 | 17
score on a scale | -1.0 (1.8) | -0.6 (1.4)

3. Secondary Outcome: Walk Distance
Description: We measured the difference in walk distance (in meters) between the first and second shuttle walk tests.
Time Frame: After the first shuttle walk test and after the second shuttle walk test
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Intervention Group (High Dose Fentanyl Sublingual Spray) | Controlled Group (Low Dose Fentanyl Sublingual Spray)
Number analyzed (Participants) | 13 | 17
meters | 43.7 [25.6 to 61.8] | 24.2 [5.8 to 42.6]

4. Secondary Outcome: Walk Time
Description: We measured the difference in walk time (in minutes) between the first and second shuttle walk tests.
Time Frame: After the first shuttle walk test and after the second shuttle walk test
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Intervention Group (High Dose Fentanyl Sublingual Spray) | Controlled Group (Low Dose Fentanyl Sublingual Spray)
Number analyzed (Participants) | 13 | 17
minutes | 0.5 [0.3 to 0.7] | 0.3 [0.18 to 0.5]

5. Secondary Outcome: Fatigue Modified Borg Score
Description: The fatigue modified Borg scale, which ranges from 0 ("none") to 10 ("worst"). We measured the change in modified fatigue Borg scale (0-10) between the first and second shuttle walk tests.
Time Frame: Before and after the first and second shuttle walk tests
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group (High Dose Fentanyl Sublingual Spray) | Controlled Group (Low Dose Fentanyl Sublingual Spray)
Number analyzed (Participants) | 13 | 17
score on a scale | -1.0 (2.8) | 0.2 (1.6)

ADVERSE EVENTS:
Time Frame: immediately before drug administration and immediately after the second walk test (approximately 20 min later)
Arm/Group | Intervention Group (High Dose Fentanyl Sublingual Spray) | Controlled Group (Low Dose Fentanyl Sublingual Spray)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/17
Other Adverse Events (participants affected / at risk) | 2/13 | 5/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (High Dose Fentanyl Sublingual Spray) (N=13) | Controlled Group (Low Dose Fentanyl Sublingual Spray) (N=17)
Dizziness (Nervous system disorders) | 1 | 5
Drowsiness (Nervous system disorders) | 2 | 1
Itchiness (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT02597478/Prot_SAP_000.pdf